CLINICAL TRIAL: NCT04795674
Title: Behavioral and Neural Target Engagement for ADHD Executive Working Memory Training
Brief Title: Target ADHD Executive Working Memory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Michael Stevens, Senior Research Scientist, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHC-2020-0305
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-02

CONDITIONS: ADHD
Keywords: Adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD EWM (Experimental): Participants will receive EWM training sessions.
  Interventions: Behavioral: EWM Training
- ADHD Placebo (Placebo Comparator): Participants will receive placebo training sessions.
  Interventions: Behavioral: Placebo Training

INTERVENTIONS:
Behavioral: EWM Training — Training tasks will target Executive Working Memory areas of the brain. Task difficulty will be adaptively increased across the 5 weeks of training based on session-to-session performance.
  Arms: ADHD EWM
Behavioral: Placebo Training — Computerized tasks with comparable engagement that do not tap executive working memory processes
  Arms: ADHD Placebo

SUMMARY:
This study will assess whether or not a novel executive working memory training intervention for Attention-Deficit/Hyperactivity Disorder can engage frontoparietal brain network treatment targets and behavioral performance.

DETAILED DESCRIPTION:
This proposal seeks support for a 2-year milestone-driven R61 initial test of target engagement in n=62 ADHD diagnosed adolescents randomized to a 'sham training' placebo or to train 4 times each week using 4 different EWM exercises that have been combined into the format of a typical cognitive training intervention. Exercise difficulty levels in the active intervention will increase across 5 weeks to continually challenge EWM ability. EWM training will use a novel, remotely-supervised 'at home' computerized training approach. If R61 EWM training target engagement milestones are met, a 3-year R33 phase will begin. The R33 will replicate target engagement in another randomized placebo-controlled trial of n=90 new ADHD adolescents and attempt to establish a convincing link between the hypothesized targets and ADHD symptom expression. It also will characterize ADHD brain activity or EWM ability changes relative to typical levels seen in an n=40 non-ADHD control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* English speaking
* Right-handed
* >5th grade reading level
* >80 IQ level

Exclusion Criteria:

* Braces, metal or implant devices
* Brain abnormality, neurological disorder
* TBI or loss of consciousness>30 minutes
* Diagnosis of Psychosis, Bipolar Disorder, ASD, PTSD, OCD, SUD, Tourette's Disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging Functional Brain Scan using a Seimens 3T Skyra. | Change in fMRI measurements from baseline assessment versus 5 weeks at the conclusion of training
  fMRI measures of brain activation and functional connectivity - Conventional measures of 'brain activation' are estimated using GLM regression models that fit the fMRI BOLD timeseries data to a model of expected hemodynamic change as elicited by fMRI versions of the executive working memory training task trials. Functional connectivity is assessed using a form of cross-correlation analysis that quantifies how much the entire BOLD timeseries in different brain regions are similar to one another. Our a priori treatment target brain regions are the superior frontal sulcus and mid-lateral prefrontal cortex region of interest. Brain activity and functional connectivity specifically to these regions represent the primary outcome measures of the study.
The experimental executive working memory training tasks | Change in scores from baseline assessment versus 5 weeks at the conclusion of training
  Will examine changes in performance accuracy on the 4 executive working memory training tasks. These are experimental, non-published tasks being tested in this project for the first time.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stevens, PhD, Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04795674/ICF_000.pdf